CLINICAL TRIAL: NCT06592820
Title: Endoscopic Ultrasound With Shear Wave Elastography for the Assessment of Liver Disease
Brief Title: Endoscopic Ultrasound Shear Wave Elastography Study
Acronym: EUS-SWE
Status: Recruiting | Type: Observational
Sponsor: Olympus Corporation of the Americas (Industry)
Responsible Party: Sponsor
Other Study IDs: 2021-GI-02
Record Dates: First submitted 2024-05-28; First posted 2024-09-19 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: MASLD; MASH; Fibrosis, Liver; Chronic Liver Disease
Keywords: Shear Wave Elastography; Shear Wave; FibroScan; Attenuation Imaging
MeSH Terms: conditions — Liver Cirrhosis | interventions — Endosonography

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- All subjects enrolled: Consecutive, eligible patients reporting for an endoscopic ultrasound liver biopsy and FibroScan for evaluation of liver fibrosis will be enrolled. EUS-SWE/ATI will be compared to liver biopsy pathology results, FibroScan (VCTE and CAP) results, and screening scores).
  Interventions: Device: Endoscopic Ultrasound Shear Wave Elastography (EUS) and Attenuation Imaging; Device: FibroScan; Device: Liver biopsy

INTERVENTIONS:
Device: Endoscopic Ultrasound Shear Wave Elastography (EUS) and Attenuation Imaging — EUS combines ultrasound technology with endoscopy to gain an internal vantage point to obtain higher resolution ultrasound images. Shear Wave is a software option on the ultrasound system EUS that provides an advanced measure and dynamic display of tissue stiffness which is being evaluated for use in assessing liver fibrosis. Attenuation Imaging (ATI) is a novel application that provides the capability to quantify and color-code the changes in attenuation coefficient of the liver that may arise with changes in liver composition (e.g., increased fat levels).
  Other Names: EUS-SWE/ATI
Device: FibroScan — A small ultrasound probe to measure the velocity of a sound wave passing through the liver. This is converted into kilopascals (kPa), which is used to assess liver fibrosis.
Device: Liver biopsy — A biopsy of liver tissue could be obtained under endoscopic ultrasound guidance, interventional radiology (percutaneously), or surgically.
  Endoscopic Ultrasound-guided liver biopsy provides high resolution images of left lobe of the liver and a good portion of the right lobe of the liver. This, coupled with Doppler capability, allows the physician to direct the biopsy needle safely into the liver for sampling under real time image guidance.
  Other Names: EUS-guided LB

SUMMARY:
This study shall be a prospective, multicenter, single arm, consecutive, interventional study conducted in a post-market setting using commercially available devices. Consecutive, eligible patients with clinical suspicion of MASLD or MASH reporting for an endoscopic ultrasound and liver biopsy for evaluation of fibrosis will be enrolled. EUS Shear Wave Elastography and Attenuation Imaging technologies will be compared to liver biopsy and FibroScan results and other non-invasive fibrosis screening modalities . The data collected during this study will be evaluated in accordance with the procedures set forth in the protocol. The main question[s] it aims to answer are:

* Establish optimal cutoffs for EUS-SWE in reference to liver biopsies staging system for liver fibrosis
* Evaluate the diagnostic performance of EUS-SWE compared to FibroScan (VCTE) and to other non-invasive fibrosis screening modalities (screening scores).

Participants will undergo:

* Endoscopic Ultrasound with Shear Wave Elastography (SWE) and Attenuation Imaging (ATI)
* Liver biopsy
* FibroScan

DETAILED DESCRIPTION:
A total of up to 300 subjects will be enrolled and treated at up to six US sites. Enrollment is expected to be completed within 18 months. Each subject will undergo procedures (EUS with SW Elastography and Attenuation Imaging, liver biopsy and FibroScan). Liver biopsy and FibroScan should be done within three months from Endoscopic ultrasound with SWE and ATI. End of study participation for a subject will be reached after pathology results have been obtained.

This study has been designed as a post-market clinical registry to evaluate the effectiveness of Endoscopic Ultrasound with Shear Wave Elastography to estimate hepatic fibrosis in patients with chronic liver disease. All consenting, eligible patients reporting for an ultrasound and liver biopsy for evaluation of fibrosis meeting the inclusion criteria will be consecutively enrolled into the study and assigned a unique study identification number.

ELIGIBILITY:
Inclusion Criteria:

1. 18 years of age or older
2. Willing and able to provide informed consent
3. Patient scheduled to undergo EUS with liver biopsy, either same session or separately; if separate, liver biopsy should be performed within 3 months of the EUS (either before or after) with no interval bariatric procedure/surgery or weight change of >10% total body weight
4. Patient scheduled to undergo or have undergone FibroScan, which should be performed within 3 months of the EUS (either before or after) with no interval bariatric procedure/surgery or weight change of >10% total body weight
5. BMI >/=28
6. Clinical suspicion of MASLD (hepatic steatosis with at least one of five cardiometabolic risk factors: 1) overweight or obesity, 2) elevated glucose, 3) low HDL-C, 4) hypertension, and/or 5) hypertriglyceridemia) or MASH (additionally characterized by the presence of inflammation and hepatocellular ballooning) with or without fibrosis, as determined by non-invasive or minimally invasive techniques (e.g. abdominal ultrasound, FibroScan)

Exclusion Criteria:

1. Patients with surgically altered anatomy that precludes adequate endosonographic visualization of the liver parenchyma
2. Prior history of Hepatitis B or C infection
3. Decompensated cirrhosis (GI bleeding, ascites, encephalopathy)
4. Histological evidence of other concomitant chronic liver disease on biopsy
5. Inadequate liver biopsy
6. Prior history of or current excess alcohol consumption (>140 g/week and >210 g/week for females and males, respectively) documented in EMR

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-09-03 (Actual); Primary Completion 2027-02-28 (Estimated); Study Completion 2027-03-28 (Estimated)

PRIMARY OUTCOMES:
Shear Wave Elastography (SWE) vs liver biopsy METAVIR staging system | During study data analysis
  Establish optimal cutoffs for EUS-SWE cutoffs in reference to liver biopsies on METAVIR staging system for significant fibrosis (F0-1 vs F2-4), advanced fibrosis (F0-2 vs F3-4), and cirrhosis (F0-3 vs F4) based on area under the receiver operator characteristics (AUROC) curve analysis.

SECONDARY OUTCOMES:
SWE vs FibroScan and other non-invasive fibrosis screening modalities ( screening scores) | During study analysis
  Evaluate the diagnostic performance of EUS-SWE compared to FibroScan (VCTE) and to other non-invasive fibrosis screening modalities (e.g., Fibrosis-4 Score (FIB-4), AST to Platelet Ratio Index (APRI), and NAFLD Fibrosis Score (NFS)).
Correlation of EUS-SWE to fibrosis staging (from liver biopsy). | During study analysis
  Evaluate the correlation of EUS-SWE to fibrosis staging (from liver biopsy).
Correlation of EUS-ATI to steatosis score (from liver biopsy) | During study analysis
  Evaluate the correlation of EUS-ATI to steatosis score (from liver biopsy).

CONTACTS AND LOCATIONS:
Overall Officials: Marvin Ryou, MD, Principal Investigator — Brigham and Women's Hospital, Boston, MA
Locations (2):
- United States (2):
  - Brigham and Women's Hospital, Boston, Massachusetts
  - Geisinger Medical Center, Danville, Pennsylvania

IPD SHARING:
Plan to Share IPD: No